CLINICAL TRIAL: NCT03090568
Title: Comparative Bioavailability Study of BIA 5-453 Under Fasted and Fed Conditions
Brief Title: Bioavailability Study of BIA 5-453
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-5453-104
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Congestive Heart Failure
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — etamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIA 5-453 Fasting (Experimental): BIA 5-453 200 mg in fasting conditions
  Interventions: Drug: BIA 5-453
- BIA 5-453 Fed (Experimental): BIA 5-453 200 mg in fed conditions
  Interventions: Drug: BIA 5-453

INTERVENTIONS:
Drug: BIA 5-453 — BIA 5-453 capsules 50 mg. Route of administration: Oral. In one period subjects received 4 capsules of 50 mg of BIA 5-453 after a fasting of at least 10 hours, and in the other period subjects were dosed with 4 capsules of 50 mg of BIA 5-453 after a standard high-fat and high-calorie meal
  Other Names: Etamicastat

SUMMARY:
The purpose of this study was to compare the bioavailability and tolerability of BIA 5-453 under fasted and fed conditions.

DETAILED DESCRIPTION:
This was a Single-centre, two-way crossover, randomised, open-label study in 12 healthy male volunteers. Subjects received a single oral 200 mg dose of BIA 5-453 following a standard meal in one period, and following at least 10 hours of fasting in another period. Treatment periods were separated by a washout interval of 2 weeks or more.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 45 years, inclusive.
* had a body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* had clinical laboratory test results clinically acceptable at screening and admission to the first treatment period.
* had negative screen for alcohol and drugs of abuse at screening and admission to the first treatment period.
* were non-smokers or smoked ≤ 10 cigarettes or equivalent per day.
* was able and willing to give written informed consent.

Exclusion Criteria:

* had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* had a clinically relevant surgical history.
* had a clinically relevant family history.
* had a history of relevant atopy or drug hypersensitivity.
* had a history of alcoholism or drug abuse.
* consumed more than 14 units of alcohol a week.
* had a significant infection or known inflammatory process at screening or admission to the first treatment period.
* had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to the first treatment period.
* used medicines within 2 weeks of admission to first period that affected the safety or other study assessments, in the investigator's opinion.
* used any investigational drug or participated in any clinical trial within 3 months prior to screening.
* participated in more than 2 clinical trials within the 12 months prior to screening.
* donated or received any blood or blood products within the 3 months prior to screening.
* was a vegetarian, vegan or with medical dietary restrictions.
* could not communicate reliably with the investigator.
* was unlikely to co-operate with the requirements of the study.
* was unwilling or unable to give written informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07-15 (Actual); Primary Completion 2008-08-14 (Actual); Study Completion 2008-08-14 (Actual)

PRIMARY OUTCOMES:
Cmax - the maximum plasma concentration | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Tmax - the time of occurrence of Cmax | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
AUC0-t - the area under the plasma concentration-time curve from time zero to the last sampling time | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
AUC0-∞ - the area under the plasma concentration versus time curve from time zero to infinity | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial's Human Pharmacology Unit, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided